CLINICAL TRIAL: NCT00664365
Title: A Single Blind, Randomised, Placebo Controlled, Single Ascending Dose Study to Evaluate the Safety, Tolerability and Pharmacokinetics of GSK958108 in Healthy Male Subjects
Brief Title: FTIH Study With GSK958108
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Purpose: Treatment
Other Study IDs: SPE111154
Record Dates: First submitted 2008-04-10; First posted 2008-04-22 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Premature Ejaculation
Keywords: Premature ejaculation.; FTIH,; GSK958108,; 5HT1a antagonist,
MeSH Terms: conditions — Premature Ejaculation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Subjects receiving GSK958108 + placebo in cohort 1 (Experimental): Eligible subjects will receive GSK958108 with a starting dose of 1 milligram. The dose escalation will be continued up to 4 ascending doses. Subjects will also receive placebo. Each treatment period will be separated by at least 7 days washout period.
  Interventions: Drug: GSK958108; Drug: Placebo
- Subjects receiving GSK958108 + placebo in cohort 2 (Experimental): Eligible subjects will start dosing once the cohort 1 has completed the treatment phase and the initial dose will be the same as top dose in Cohort1.The dose escalation will be continued up to 4 ascending doses. Subjects will also receive placebo. Each treatment period will be separated by at least 7 days washout period.
  Interventions: Drug: GSK958108; Drug: Placebo

INTERVENTIONS:
Drug: GSK958108 — GSK958108 oral tablets will be available with dosing strengths of 1 milligram, 5 milligrams, 25 milligrams and 50 milligrams. It will be a brownish-yellow film coated round shape tablet. The tablets have to be swallowed completely with 240 milliliters of water, without chewing over a period of five minutes.
Drug: Placebo — Placebo tablets will be brownish-yellow film coated round shape tablets, administered orally. The tablets have to be swallowed completely with 240 milliliters of water, without chewing over a period of five minutes.

SUMMARY:
This study is the first administration of GSK958108 to man. The study will evaluate the safety, tolerability and pharmacokinetics of single ascending doses of GSK958108 and evaluate the effect of food on GSK958108 pharmacokinetics

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Male between 18 and 65 years of age
* Male subjects must agree to use one of the contraception methods as per protocol. This criterion must be followed from the time of the first dose of study medication until 3 months after last dose.
* Body weight > 50 kg (110 lbs) for men and BMI within the range 19.0 - 29.9 kg/m2 inclusive)
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* The subject has a visual acuity that is equivalent to 20/20 in each eye, with appropriate correction if needed
* The subject is able to cooperate in all part of the eye examination (including dilation with mydriatics)

Exclusion Criteria:

* The subject has a positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines (Can be repeated once at screening).
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening (with the exception of phase I hepatic impairment studies, oncology studies, hepatitis, hepatic fibrosis, or HIV studies).
* A positive test for HIV antibody.
* History of long QT syndrome (personal or family) or other cardiac conduction disorder, or other clinically significant cardiac disease.
* The subject has prolactin, total and free testosterone, LH, FSH outside of the normal range (to be discussed with the Medical Monitor, if necessary).
* History of regular alcohol consumption within 6 months of the study defined as:

  - an average weekly intake of greater than 21 units or an average daily intake of greater than 3 units (males). One unit is equivalent to a half-pint (220mL) of beer or 1 (25ml) measure of spirits or 1 glass (125ml) of wine.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity or intolerance to drugs that effect serotonin, including serotonin-reuptake inhibitors (SSRIs),or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* The subject has a history of migraine.
* The subject has a history of psychiatric illness.
* Any history of suicidal attempts or behaviour.
* The subject has a history of any eye disorder or is color blind, excluding myopia and presbyopia.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice [and/or pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices] from 7 days prior to the first dose of study medication.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2008-04-12 (Actual); Primary Completion 2008-08-22 (Actual); Study Completion 2008-08-22 (Actual)

PRIMARY OUTCOMES:
Safety will be evaluated by adverse event monitoring, physical and neurological examination, pupil size, Eye assessment; 12-lead ECG, vital signs and laboratory parameters. These assessments will be conducted at several timepoints after each dosing. | Up to Day 19

SECONDARY OUTCOMES:
To assess the food effect on the pharmacokinetics of GSK958108 in healthy male volunteers | Up to Day 5

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom

REFERENCES:
- See also: Results for study SPE111154 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/SPE111154?search=study&study_ids=SPE111154#rs